CLINICAL TRIAL: NCT02010931
Title: A Retrospective Analysis of Hematological Relapse Free Survival and Overall Survival in Adult Patients With Philadelphia-Negative B-Precursor Acute Lymphoblastic Leukemia in Complete Hematological Remission With Minimal Residual Disease
Brief Title: Retrospective Analysis of Survival in Adult MRD Positive Acute Lymphoblastic Leukemia Patients
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Collaborators: European EWALL study groups (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20120148
Record Dates: First submitted 2013-11-25; First posted 2013-12-13 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- primary: subjects who are 18 years or older, who have minimal residual disease detected by PCR at a level of 1/10-3 or higher, who are free form allogeneic stem cell transplantation until hematological relapse or until 18 months after minimal residual disease detection (whichever comes first)

SUMMARY:
A retrospective analysis of historical data looking at relapse free survival and overall survival rates in adult philadelphia negative B-pre-cursor acute lymphoblastic leukemia patients.

DETAILED DESCRIPTION:
A retrospective observational study reviewing historical survival data (relapse free survival and overall survival) for adult patients who have philadelphia negative B-precursor acute lymphoblastic leukemia, and are in complete hematological remission with minimal residual disease.

ELIGIBILITY:
Inclusion Criteria:

* patients with Philadelphia-negative B-Precursor Acute Lyphmoblastic Leukemia in complete hematological remission defined as less than 5% blasts in bone marrow after at least 3 intensive chemotherapy blocks (i.e. any standard or investigational regimen according to adult protocols as long as 3 age appropriate chemotherapy blocks were given, this also includes relapse treatment
* detection of minimal residual disease (molecular failure or molecular relapse) at a level of greater than or equal to 10*(-4) by PCR or greater than or equal to 10*(-3) by flow cytometry at a reference lab
* Age 15 or greater at time of initial diagnosis with acute lymphoblastic leukemia. For patients aged 15-17 treatment according to adult protocols is required
* Initial diagnosis in the year 2000 or later
* History of acute lymphoblastic leukemia treatment (including response to first therapy, number of prior relapses) is available
* Relapse status and disease follow up after timepoint of minimal residual disease detection is available

Exclusion Criteria:

* Patients with extramedullary disease at timepoint of minimal residual disease detection
* Use of Blinatumomab within 18 months of minimal residual disease detection
* Allogeneic hematopoietic stem cell transplantation prior to minimal residual disease detection at the required level

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
hematological relapse free survival | Approximately 18 months
  to estimate the hematological relapse free survival in patients who are 18 years or older, who have minimal residual disease detected by PCR at a level of 1/10-3 or higher, who are free form allogeneic stem cell transplantation until hematological relapse or until 18 months after minimal residual disease detection (whichever comes first)

SECONDARY OUTCOMES:
hematological relapse free survival | Approximately 18 months
  to estimate the hematological relapse free survival in patients who are 15 years or older, who have minimal residual disease regardless of detection method, with or without stem cell transplantation within18 months of minimal residual disease detection
overall survival | Approximately 18 months
  to estimate overall survival in the 2 sets of patients described in the primary outcome measure, and the first secondary outcome measure.
mortality rate | 100 days following allogeniec stem cell transplantation
  to estimate the mortality rate (proportion) at 100 days following allogeneic stem cell transplantation in patients who received an allogeneic stem cell transplantation within 18 months after minimal residual disease detection

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- Research Site, Brno, Czechia
- Research Site, Paris, France
- Research Site, Frankfurt am Main, Germany
- Italy (3):
  - Research Site, Bologna
  - Research Site, Roma
  - Research Site, Venezia
- Research Site, Gliwice, Poland
- Research Site, Moscow, Russia
- Research Site, Badalona, Catalonia, Spain
- Research Site, London, United Kingdom

REFERENCES:
- [Background] Gokbuget N, Dombret H, Giebel S, Bruggemann M, Doubek M, Foa R, Hoelzer D, Kim C, Martinelli G, Parovichnikova E, Maria Ribera J, Schoonen M, Tuglus C, Zugmaier G, Bassan R. Blinatumomab vs historic standard-of-care treatment for minimal residual disease in adults with B-cell precursor acute lymphoblastic leukaemia. Eur J Haematol. 2020 Apr;104(4):299-309. doi: 10.1111/ejh.13375. Epub 2020 Jan 24. PMID 31876009
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com